CLINICAL TRIAL: NCT03347552
Title: Home-Based Mental Health Evaluation (HOME): A Multi-Site Trial
Brief Title: Home-Based Mental Health Evaluation (HOME)
Acronym: HOME
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 13-2982
Record Dates: First submitted 2017-11-15; First posted 2017-11-20 (Actual); Last update posted 2018-04-17 (Actual); Status verified 2018-04

CONDITIONS: Suicide and Self-harm
Keywords: treatment engagement
MeSH Terms: conditions — Suicide; Self-Injurious Behavior

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The blind assessor will administer follow up measures. In order to keep the assessor blind to participant status (active vs. control), research staff will facilitate phone calls. To monitor blinding, the blind assessor will record if participants inadvertently un-blind themselves during the assessment and also record their guess to which treatment condition (active versus E-CARE)participants were allocated.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Treatment (Experimental): Participants in the active arm will be enrolled in the HOME Program.
  Interventions: Behavioral: HOME
- E-CARE (No Intervention): Receiving enhanced care as usual. Participants at these sites are described as receiving "enhanced care as usual" or "E-CARE" because they will be recruited, enrolled and complete baseline and follow-up assessments in addition to care as usual.

INTERVENTIONS:
Behavioral: HOME — Prior to discharge from the inpatient unit, the HOME program provider or another member of the research team, will meet individually with the Veteran to provide further information regarding the HOME program intervention. Efforts are made to schedule the initial phone call and home visit that occur during the first week after discharge. Following the home visit, the HOME provider may continue to have weekly contact with the Veteran via the telephone or in person until he or she is disenrolled following engagement in outpatient care. "Engaged in care" is defined as attendance at two individual outpatient mental health appointments or engagement in equivalent or elevated care as determined by the PI. All clinical contacts with the Veteran may include the following: suicide risk assessment, review and modification of the Veteran's safety plan, review and modification of the discharge plan, involvement of the Veteran's support system, and facilitation of engagement in outpatient care.
  Arms: Active Treatment

SUMMARY:
The purpose of this project is to investigate the effectiveness of the Home-Based Mental Health Evaluation (HOME) program, which is an innovative and culturally-relevant suicide prevention intervention for Veterans aimed at increasing treatment engagement and decreasing suicide risk following psychiatric hospitalization, a period of heightened suicide risk.

DETAILED DESCRIPTION:
The purpose of this project is to investigate the effectiveness of the Home-Based Mental Health Evaluation (HOME) program, which is an innovative and culturally-relevant suicide prevention intervention for Veterans aimed at increasing treatment engagement and decreasing suicide risk following psychiatric hospitalization, a period of heightened suicide risk. The research project employs a multi-site two-arm interventional trial design to study the effectiveness of the HOME program. Effectiveness of the treatment will be evaluated by comparing Veterans receiving the HOME program at two active treatment sites, Denver and Philadelphia Department of Veterans Affairs Medical Centers (VAMCs), to with those receiving care at two control sites, Houston and Portland VAMCs. The current protocol describes procedures as they will occur at all sites, including those completed locally at the Denver VAMC, which is the lead site for the study.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18-89
2. Able to provide a phone number and the location of a residence at which they can be reached
3. Planned location of discharge is a safe environment for the HOME provider to visit*
4. Agree to receive the HOME program intervention (active site participants only)
5. Ability to adequately respond to questions regarding the informed consent procedure

Exclusion Criteria:

1. Receiving services from the Mental Health Intensive Case Management (MHICM) or Domiciliary program or being directly transferred to further inpatient or residential treatment
2. Enrolled in other intervention studies that may affect the outcome of this study, or where this study may affect the outcome of the other study, until the subject has completed their participation in the other study
3. Current involvement in the criminal justice system as a prisoner or ward of the state.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 323 (Actual)
Dates: Start 2014-04-29 (Actual); Primary Completion 2016-09-01 (Actual); Study Completion 2016-11-30 (Actual)

PRIMARY OUTCOMES:
Treatment Engagement 1 | From discharge from the hospital through 90 days post discharge
  Access to participants' VA electronic medical record will be utilized to address the hypothesis that Veterans participating in the HOME program will be significantly more likely to engage in treatment and or care more quickly. Data collection may be facilitated by VA's Compensation and Pension Record Interchange (CAPRI) and VA's Corporate Data Warehouse (CDW).
Treatment Engagement 3 | From discharge from the hospital through 90 days post discharge
  Access to participants' VA electronic medical record will be utilized to address the hypothesis that Veterans participating in the HOME program will be significantly more likely to attend more outpatient appointments. Data collection may be facilitated by VA's Compensation and Pension Record Interchange (CAPRI) and VA's Corporate Data Warehouse (CDW).

SECONDARY OUTCOMES:
Lower Suicidal Ideation scores | 3 months post-discharge
  Compared to the E-CARE group, Veterans participating in the HOME program will report significantly lower suicidal ideation scores on the Scale for Suicidal Ideation. The Scale for Suicidal Ideation (SSI) will be used to measure this outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Bridget B Matarazzo, PsyD, Principal Investigator — VA Rocky Mountain MIRECC
Locations (3):
- United States (3):
  - VA Portland Health Care System, Portland, Oregon
  - Philadelphia VA Medical Center, Philadelphia, Pennsylvania
  - Michael E. DeBakey VA Medical Center, Houston, Texas

REFERENCES:
- [Derived] Matarazzo BB, Gerard GR, Jankovsky MC, Oslin DW, Brenner LA. Feasibility and Acceptability of the HOME Program for Veterans Recently Discharged from a Psychiatric Hospitalization. Adm Policy Ment Health. 2021 Nov;48(6):974-982. doi: 10.1007/s10488-021-01109-7. Epub 2021 Feb 1. PMID 33523330